CLINICAL TRIAL: NCT02097485
Title: A Randomised, Double-Blind, Vehicle-Controlled Study of Ovicidal Efficacy and Safety of Abametapir 0.74% Administered for the Treatment of Head Lice Infestation
Brief Title: Ovicidal Efficacy and Safety of Abametapir Lotion 0.74% Administered for the Treatment of Head Lice Infestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ha03-008
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Head Lice Infestation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abametapir Lotion 0.74% w/w (Active Comparator): Topically administered to hair and scalp for 10 minutes application.
  Interventions: Drug: Abametapir Lotion 0.74% w/w
- Vehicle Lotion (Placebo Comparator): Administered to scalp and hair for 10 minutes application.
  Interventions: Drug: Vehicle Lotion

INTERVENTIONS:
Drug: Abametapir Lotion 0.74% w/w — 200mL abametapir lotion topically administered to the scalp and hair and once fully saturated left for 10 minutes and then washed out thoroughly with warm water.
  Arms: Abametapir Lotion 0.74% w/w
Drug: Vehicle Lotion — control to abametapir: 200mL Vehicle Lotion topically administered to the scalp and hair and once fully saturated left for 10 minutes and then washed out thoroughly with warm water.
  Arms: Vehicle Lotion

SUMMARY:
The purpose of the study was to evaluate ovicidal efficacy of a single application of abametapir lotion 0.74% w/w intended for the treatment of head lice.

DETAILED DESCRIPTION:
This was a double-blind, randomised, vehicle-controlled, parallel group study in males and females, aged three years and older with active head lice infestation. The study was designed to assess the ovicidal efficacy of a single application of abametapir lotion 0.74% w/w compared to a vehicle control, when applied to the scalp and hair for 10 minutes at the study site. This study used an ex vivo method of assessment for ovicidal efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female based on medical history
2. Six months of age or older.
3. Has an active head lice infestation with a minimum of 3 live head lice and at least 10 undamaged and unhatched head lice eggs in their hair.
4. Agrees to an examination for head lice and compliance with the study procedures.
5. All adult subjects must sign a written voluntary informed consent. For minors, the parent/ legal guardian agrees to the subject participating in the study as determined by the signing of an assent of informed consent.

Exclusion Criteria:

1. Has scalp disease or a history of allergies or prior reactions to any head lice products.
2. Has a condition that, in the opinion of the Investigator, may interfere with the study.
3. Is receiving systemic or topical medication, which in the opinion of the Investigator, may compromise the integrity of the safety and/or efficacy assessments.
4. Had treatment (over-the-counter (OTC) or home remedy medication) for head lice within 14 days prior to Day 0.
5. Has received an investigational agent within 30 days prior to Day 0.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Arnold, MBBS, Principal Investigator — National Head Lice Treatment Centre, Ringwood East, Victoria, Australia, 3135
Locations (1):
- National Head Lice Treatment Centre, Ringwood East, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Population included subjects who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (3.43) | 8.3 (2.95) | 8.5 (3.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 25 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Hatched Eggs Pre Treatment Relative to Post Treatment
Description: Percentage of hatched eggs pre treatment relative to percentage of hatched eggs post treatment for the abametapir and vehicle treated eggs following 14 day incubation. The difference between post treatment percent hatching and pre-treatment percent hatching was calculated i.e. post-treatment minus pre-treatment hatching percent.
Time Frame: 14 days
Population: Full Analysis Set (FAS) included all randomized subjects who received any amount of study treatment and had at least 1 viable pre-treatment egg and 1 viable post-treatment egg evaluable for analysis.
Measure: Mean (95% Confidence Interval); unit: Percent hatched eggs post versus pre Rx
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion
Number analyzed (Participants) | 25 | 25
Percent hatched eggs post versus pre Rx | -92.9 [-99.4 to -86.5] | -42.3 [-54.4 to -30.2]

ADVERSE EVENTS:
Time Frame: AEs were collected from the start of treatment on Day 0 through the Day 7 follow up visit (Approximately 8 days).
Arm/Group | Abametapir Lotion 0.74% w/w | Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 4/25 | 2/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abametapir Lotion 0.74% w/w (N=25) | Vehicle Lotion (N=25)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No